CLINICAL TRIAL: NCT02984137
Title: A Prospective Longitudinal Neuroimaging and Biomarker Cohort Study in Idiopathic Rapid Eye Movement(REM) Sleep Behavior Disorder
Brief Title: Prospective Neuroimaging Investigation of Idiopathic REM Sleep Behavior Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jee-Young Lee, Associate Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 16-2013-101
Record Dates: First submitted 2016-11-30; First posted 2016-12-06 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Parkinson Disease; REM Sleep Behavior Disorder
Keywords: Lewy body disease; REM Sleep Behavior Disorder; Parkinson disease; Imaging; Bio-markers; Prospective cohort
MeSH Terms: conditions — Parkinson Disease; REM Sleep Behavior Disorder; Lewy Body Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- idiopathic RBD group (Experimental): A group of patients diagnosed as idiopathic RBD that is confirmed by polysomnography. Interventions as testing, evaluation, samplings at baseline, then repeat at 2 years and 4 years of prospective follow-up. thereafter only clinical observations until Lewy body disease is diagnosed.
  Interventions: Other: testing, evaluation, sampling
- incident PD group (Active Comparator): A group of patients who are newly diagnosed as Parkinson's disease, and never been treated with prolonged history of probable RBD. Interventions as testing, evaluation, sampling at baseline and then evaluations only at 3 year follow-up after anti-parkinsonian treatment.
  Interventions: Other: testing, evaluation, sampling
- Control (Placebo Comparator): Control group includes elderly controls without neurodegerative diseases examined by neurologists. Interventions as testing, evaluation, sampling at baseline only.
  Interventions: Other: testing, evaluation, sampling

INTERVENTIONS:
Other: testing, evaluation, sampling — neuroimaging biomarkers using positron emission tomography and magnetic resonance imaging, and evaluation of neurological & neurocognitive status by using a predefined neuropsychological assessment battery.

SUMMARY:
This is a prospective cohort study to evaluate degenerative changes in the brain by performing functional imaging analysis in patients with RBD and its correlations with clinical symptoms and dopaminergic degeneration. This study also evaluates cognitive changes with functional imaging measures and olfactory and other premotor symptoms of Lewy body disease. This study also collects gene extracts and sera to develop a biomarker for early detection of neurodegeneration.

DETAILED DESCRIPTION:
This study will include 3 groups in relation with RBD: idiopathic RBD (iRBD), PD- RBD, normal controls without RBD. In all groups, neurological examinations, olfactory testings, nonmotor symptoms evaluations, neuropsychological evaluations (detailed outcomes are in the outcome section) will be performed at baseline evaluation after enrollment. Image data will be obtained on following modalities: brain magnetic resonance imaging (MRI), 18F-N-ω-fluoropropyl- 2β-carbomethoxy- 3β-(4-iodophenyl) nortropane ([18F]FP-CIT) positron emission tomography (PET), and 18F-fludeoxyglucose([18F]FDG) PET.

To assess progression toward Lewy body disorders, patients in iRBD group will be evaluated at 2, and 4 years of follow-up visit. Clinical, neuropsychological tests, brain MRI, and two PET scans will be administered. After 4 years, patients who are willing to participate will be additionally followed-up yearly as a routine clinical visit with clinical and neurological examinations until obvious signs of Lewy body diseases will develop.

In PD-RBD group, patients will be evaluated at 3-year follow-up period amongst days of routine clinic visits with administering clinical and neuropsychological tests.

ELIGIBILITY:
Inclusion Criteria:

iRBD group:

* A diagnosis of RBD according to the international classification of sleep disorders-2 (ICSD-2) criteria
* No current neurological diseases related with RBD
* Male or female aged from 30 to 80 years old at screening
* Subject enrolled voluntarily and understood the contents of the study

PD group:

* A diagnosis of PD according to the UK Brain Bank Diagnostic Criteria
* A diagnosis of RBD according to the international classification of sleep disorders-2 (ICSD-2) criteria
* Male or female aged from 30 to 80 years old at screening
* Subject enrolled voluntarily and understood the contents of the study

Control group:

* No current neurological or psychiatric diseases related with RBD
* Male or female aged from 30 to 80 years old at screening
* Age and sex matched with those of subjects in iRBD group
* Subject enrolled voluntarily and understood the contents of the study

Exclusion Criteria:

* Clinically significant cognitive decline unable to follow the study (Mini-mental state examination [MMSE] score less than 20)
* History of psychiatric illnesses (ex. depression)
* Unable to walk and cooperate to the examination
* Unable to take magnetic resonance imaging or positron emission tomography
* Existence of illness or problems which makes difficult to be enrolled to the study judged by clinicians

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Frequency of development of Lewy body diseases | up to 4-years follow-up
  idiopathic RBD group only

SECONDARY OUTCOMES:
Parkinsonian motor symptoms score change measured by the unified Parkinson's disease rating scale (MDS-UPDRS) | from baseline to 2-years and 4-years follow-up (iRBD group), to 3-years follow-up (PD-RBD group)
  descriptive, intragroup analysis
Nonmotor symptoms profile change assessed by a combined evaluatin using the non-motor symptom scale and part I of the MDS-UPDRS | from baseline to 2-years and 4-years follow-up (iRBD group), to 3-years follow-up (PD-RBD group)
  descriptive, intragroup analysis
Cognitive change measured by the neuropsychological test battery | from baseline to 2-years ad 4-years follow-up (iRBD group), to 3-years follow-up (PD-RBD group)
  descriptive, intragroup analysis
Degenerative brain changes predicted by MRI (diffusion tensor analysis and volumetry) | from baseline to 2-years and 4-years follow-up (iRBD group only)
  descriptive, intragroup analysis
Functional network changes predicted by the resting-state functional MRI | from baseline to 2-years and 4-years follow-up (iRBD group only)
  descriptive, intragroup analysis
Degenerative brain changes predicted by [18F]FP-CIT PET | from baseline to 2-years and 4-years follow-up (iRBD group only)
  descriptive, intragroup analysis
Functional network changes predicted by [18F]FDG PET | from baseline to 2-years and 4-years follow-up (iRBD group only)
  descriptive, intragroup analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jee-Young Lee, MD, PhD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided